CLINICAL TRIAL: NCT02948673
Title: The Production of Reactive Oxygen Species in Response to Glutathione Supplementation and Acute Exercise in Patients With Type 2 Diabetes
Brief Title: The Production of Reactive Oxygen Species in Response to Glutathione Supplementation and Acute Exercise
Acronym: DIMITOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Steen Larsen, Assistant Professor, DMSci., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DIMITOS
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes; Oxidative Stress; Mitochondrial Reactive Oxygen Species Production
Keywords: type 2 diabetes; mitochondrial reactive oxygen species production; oxidative stress; antioxidant treatment; glutathione supplementation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): 4 placebo tablets/day (2 in the morning and 2 in the evening)
  Interventions: Other: Placebo
- Glutathione (Active Comparator): 4 oral GSH tablets/day (2 in the morning and 2 in the evening)
  Interventions: Dietary Supplement: Glutathione

INTERVENTIONS:
Dietary Supplement: Glutathione — 4 oral GSH tablets/day (1000mg/day) for 4 weeks
  Other Names: Setria Glutathion
  Arms: Glutathione
Other: Placebo — 4 oral placebo tablets for 4 weeks
  Arms: Control

SUMMARY:
Objectives: The research focus of the study is the production of reactive oxygen species (ROS) in patients with type 2 diabetes (T2D) in response to glutathione (GSH) supplementation and in response to acute exercise.

Oxidative stress is suggested as a possible causative factor in the pathophysiology of skeletal muscle insulin resistance. GSH is the most abundant endogenous antioxidant in the cell and thus, a crucial protector against oxidative stress and insulin resistance. It has been found that patients with T2D have a decreased level of GSH in plasma and that 1 h GSH infusion improves skeletal muscle glucose uptake by ~25% and the redox environment in patients with T2D. Therefore, we want to investigate the effect of 3 months of GSH supplementation on skeletal muscle insulin sensitivity and mitochondrial ROS production in patients with T2D and healthy controls.

Hypothesis: Oral GSH supplementation will improve skeletal muscle insulin sensitivity in patients with T2D and this effect will be linked to a reduced mitochondrial ROS production in the skeletal muscle.

In contrast to the link between oxidative stress and insulin resistance, ROS produced in response to exercise is an important physiological stimulus as it is suggested to play a key role in the beneficial mitochondrial biogenesis observed in response to training. It has been reported that some patients with T2D have a diminished mitochondrial biogenesis in response to training, but the reason for this defect is not known. We want to investigate the link between exercise-stimulated ROS production and the mitochondrial biogenesis response in patients with T2D and healthy controls in response to acute exercise at two different intensities.

Hypothesis: Considering the pathological condition of T2D skeletal muscle (i.e. high chronic ROS level), we speculate that a lower exercise intensity, leading to a lower exercise-stimulated ROS production is a more optimal stimulus (i.e. not to high) for mitochondrial biogenesis in patients with T2D.

DETAILED DESCRIPTION:
ROS production in response to glutathione supplementation:

Today, 387 million people worldwide suffer from T2D and this number is expected to increase to 592 million in 2035. Skeletal muscle is responsible for ~75% of the total glucose uptake, making skeletal muscle the quantitatively most important tissue when it comes to insulin resistance (1). It has been suggested that oxidative stress may represent a possible causative factor in the pathophysiology of skeletal muscle insulin resistance. The link between ROS and skeletal muscle insulin resistance has been established both in vitro and in vivo (2, 3), but few studies have actually measured ROS production in skeletal muscle of T2D patients (4-6). Mitochondria are a source of ROS, and also a major target of oxidative damage (7). The mitochondrial defense system against oxidative stress relies on endogenous antioxidants. Glutathione (GSH) is the most abundant endogenous antioxidant in the cell and thus, a crucial protector against oxidative stress and insulin resistance (8). Supporting this, patients with T2D have a decreased level of GSH and an increased level of oxidized GSH (GSSG) in plasma (9) and insulin resistant subjects are reported to have an increased mitochondrial ROS production as well as a reduced GSH/GSSG ratio in skeletal muscle compared to healthy controls (3). In addition, 1 h glutathione infusion has been found to increase glucose uptake in patients with T2D by ~25% and to improve the redox environment, as reflected by an increased GSH/GSSG ratio in plasma; effects that were not seen in the healthy controls (10). The effect of prolonged oral GSH supplementation on skeletal muscle insulin sensitivity and mitochondrial ROS production in patients with T2D has, to our knowledge, never been investigated.

Research questions 1: Does oral GSH supplementation improve skeletal muscle insulin sensitivity in patients with T2D and healthy controls? And if so, can this effect be linked to a more beneficial redox state in the muscle cell? Hypothesis: Oral GSH supplementation will improve skeletal muscle insulin sensitivity in patients with T2D and this effect will be linked to a reduced mitochondrial ROS production in the skeletal muscle.

ROS production in response to acute exercise:

Acute exercise induces a marked increase in the transcription of peroxisome proliferator-activated receptor-γ coactivator-1α (PGC-1α) (11), and therefore, PGC-1α is believed to play a key role in training-induced mitochondrial biogenesis (12). Contraction of rat skeletal muscle cells increases ROS production and PGC-1α mRNA expression, but in the presence of antioxidants, ROS production is reduced and the increase in PGC-1α mRNA is abolished (13). Also, exercise combined with allopurinol (an inhibitor of ROS production) severely attenuates the magnitude of the exercise-induced increased PGC-1α mRNA in rats, compared to exercise alone (14). These findings suggest that PGC-1α, at least in part, is regulated through a mechanism that involves ROS. Furthermore, it has been suggested that ROS regulates PGC-1α via activation of AMP-activated protein kinase (AMPK) (15). Interestingly, subjects with insulin resistance have a decreased exercise-stimulated AMPK activity, compared to lean controls (16, 17), which might explain the attenuated training-induced mitochondrial biogenesis observed in some patients with T2D (5, 17, 18), but not all (19). Whether ROS production is implicated in an abnormal training response is not known. Our current knowledge of ROS in response to acute exercise is derived from studies in animals and cells, and no study has, to our knowledge, investigated the link between ROS and mitochondrial biogenesis in patients with T2D in response to acute exercise.

Research questions 2: Does the exercise-induced increased ROS production required for a mitochondrial biogenesis response differ between patients with T2D and healthy controls? If so, does low intensity exercise reduce the transient ROS production and thus, result in a higher mitochondrial biogenesis response in patients with T2D, compared to exercise at high intensity? Hypothesis: Considering the pathological condition of T2D skeletal muscle (i.e. high chronic ROS level), it is hypothesized that a lower exercise intensity, leading to a lower exercise-stimulated ROS production is a more optimal stimulus (i.e. not to high) for mitochondrial biogenesis in patients with T2D.

Material and methodology:

20 patients with T2D (non-insulin dependent) and 20 healthy controls will be recruited to the study. The two groups will be matched on age, weight and maximal oxygen consumption (VO2 max).

Approach for the study: The study is a double blinded randomized placebo controlled trial.

At each attendance to the laboratory (except for the day of screening), the subjects are asked to:

* Report to the laboratory in an overnight fasted state
* Abstain from alcohol and physical activity 24 hours prior to each study day.
* Repeat the same diet as the enclosed 24-hour recall questionnaire prescribes (the subjects are also asked to complete a 24-hour dietary recall questionnaire on their first attendance to the laboratory)

Screening: Before the subjects are included in the study, a standard clinical examination will be conducted, including medical history, glycated hemoglobin (HbA1c) and ECG.

If included in the study, the subjects undergoes 3 experimental days before and after the intervention.

Test day 1:

* Dual Energy X-ray Absorptiometry-scan to measure body composition,
* Incremental exercise test to determine the exercise intensity that elicits maximal fat oxidation (Fatmax test)
* Incremental exercise test to exhaustion to determine VO2 max.

Test day 2:

* Muscle biopsies from vastus lateralis (basal, immediately after exercise cessation and after 90 min of recovery)
* Acute exercise tests on bicycle ergometers at 70% of VO2 max (moderate intensity) or at 50% of VO2 max (low intensity). The two exercise tests will be matched for total amount of work (kJ).

  10 subjects with T2D and 10 control subjects are randomized to each exercise test.

Test day 3:

* Measurement of resting metabolic rate by canopy hood (basal and during the clamp)
* Intravenous glucose tolerance test
* Hyperinsulinaemic euglycaemic clamp

After the experimental days, the subjects are randomized into placebo or GSH supplementation and instructed to consume either 1000 mg GSH/day or placebo daily (2 tablets in the morning and 2 tablets in the evening) for 4 weeks.

Statistical considerations:

The comparison of the groups or the interventions will be performed using a one-way or a two-way ANOVA test with repeated measures, as appropriate. Based on the variation shown in previous studies an expected 80% power and a significance level of P<0.05, power calculations have shown that 12 subjects in each group is sufficient in regards to mitochondrial functionality measurements and insulin sensitivity. Data from a previous study investigating GSH in healthy subjects indicates that 15 subjects are needed in order to find a difference in this parameter (3).

ELIGIBILITY:
Inclusion Criteria:

For patients with type 2 diabetes:

* Male
* 30-50 years
* BMI: 28-35
* ECG with no evidence of heart disease
* HbA1c > 6.5% (48mmol/mol)

For control subjects:

* Male
* 30-50 years
* BMI: 28-35
* ECG with no evidence of Heart disease

Exclusion Criteria:

For patients with type 2 diabetes::

* Insulin treatment
* Antioxidant supplementation or other dietary supplements
* Cholesterol lowering medicine

For control subjects:

* Antioxidant supplementation or other dietary supplements
* Cholesterol lowering medicine

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12 weeks
  Difference in insulin sensitivity (measured as glucose infusion rate during a hyperinsulinaemic euglycaemic clamp) between patients with type 2 diabetes receiving glutathione supplementation and patients with type 2 diabetes receiving placebo.

SECONDARY OUTCOMES:
Mitochondrial reactive oxygen species production | 12 weeks
  Difference in the mitochondrial reactive oxygen species production between patients with type 2 diabetes receiving glutathione supplementation and patients with type 2 diabetes receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Steen Larsen, Ass. prof., Principal Investigator — University of Copenhagen
Locations (1):
- Xlab, Department of Biomedical Sciences, Faculty Of Health Sciences, University of Copenhagen, Copenhagen, Nørrebro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFronzo RA. Lilly lecture 1987. The triumvirate: beta-cell, muscle, liver. A collusion responsible for NIDDM. Diabetes. 1988 Jun;37(6):667-87. doi: 10.2337/diab.37.6.667. No abstract available. PMID 3289989
- [Background] Houstis N, Rosen ED, Lander ES. Reactive oxygen species have a causal role in multiple forms of insulin resistance. Nature. 2006 Apr 13;440(7086):944-8. doi: 10.1038/nature04634. PMID 16612386
- [Background] Anderson EJ, Lustig ME, Boyle KE, Woodlief TL, Kane DA, Lin CT, Price JW 3rd, Kang L, Rabinovitch PS, Szeto HH, Houmard JA, Cortright RN, Wasserman DH, Neufer PD. Mitochondrial H2O2 emission and cellular redox state link excess fat intake to insulin resistance in both rodents and humans. J Clin Invest. 2009 Mar;119(3):573-81. doi: 10.1172/JCI37048. Epub 2009 Feb 2. PMID 19188683
- [Background] Abdul-Ghani MA, Jani R, Chavez A, Molina-Carrion M, Tripathy D, Defronzo RA. Mitochondrial reactive oxygen species generation in obese non-diabetic and type 2 diabetic participants. Diabetologia. 2009 Apr;52(4):574-82. doi: 10.1007/s00125-009-1264-4. Epub 2009 Jan 30. PMID 19183935
- [Background] Hey-Mogensen M, Hojlund K, Vind BF, Wang L, Dela F, Beck-Nielsen H, Fernstrom M, Sahlin K. Effect of physical training on mitochondrial respiration and reactive oxygen species release in skeletal muscle in patients with obesity and type 2 diabetes. Diabetologia. 2010 Sep;53(9):1976-85. doi: 10.1007/s00125-010-1813-x. Epub 2010 Jun 6. PMID 20526759
- [Background] Chanseaume E, Barquissau V, Salles J, Aucouturier J, Patrac V, Giraudet C, Gryson C, Duche P, Boirie Y, Chardigny JM, Morio B. Muscle mitochondrial oxidative phosphorylation activity, but not content, is altered with abdominal obesity in sedentary men: synergism with changes in insulin sensitivity. J Clin Endocrinol Metab. 2010 Jun;95(6):2948-56. doi: 10.1210/jc.2009-1938. Epub 2010 Apr 9. PMID 20382691
- [Background] Murphy MP. How mitochondria produce reactive oxygen species. Biochem J. 2009 Jan 1;417(1):1-13. doi: 10.1042/BJ20081386. PMID 19061483
- [Background] Richie JP Jr, Nichenametla S, Neidig W, Calcagnotto A, Haley JS, Schell TD, Muscat JE. Randomized controlled trial of oral glutathione supplementation on body stores of glutathione. Eur J Nutr. 2015 Mar;54(2):251-63. doi: 10.1007/s00394-014-0706-z. Epub 2014 May 5. PMID 24791752
- [Background] Calabrese V, Cornelius C, Leso V, Trovato-Salinaro A, Ventimiglia B, Cavallaro M, Scuto M, Rizza S, Zanoli L, Neri S, Castellino P. Oxidative stress, glutathione status, sirtuin and cellular stress response in type 2 diabetes. Biochim Biophys Acta. 2012 May;1822(5):729-36. doi: 10.1016/j.bbadis.2011.12.003. Epub 2011 Dec 11. PMID 22186191
- [Background] De Mattia G, Bravi MC, Laurenti O, Cassone-Faldetta M, Armiento A, Ferri C, Balsano F. Influence of reduced glutathione infusion on glucose metabolism in patients with non-insulin-dependent diabetes mellitus. Metabolism. 1998 Aug;47(8):993-7. doi: 10.1016/s0026-0495(98)90357-2. PMID 9711998
- [Background] Pilegaard H, Saltin B, Neufer PD. Exercise induces transient transcriptional activation of the PGC-1alpha gene in human skeletal muscle. J Physiol. 2003 Feb 1;546(Pt 3):851-8. doi: 10.1113/jphysiol.2002.034850. PMID 12563009
- [Background] Hood DA. Invited Review: contractile activity-induced mitochondrial biogenesis in skeletal muscle. J Appl Physiol (1985). 2001 Mar;90(3):1137-57. doi: 10.1152/jappl.2001.90.3.1137. PMID 11181630
- [Background] Silveira LR, Pilegaard H, Kusuhara K, Curi R, Hellsten Y. The contraction induced increase in gene expression of peroxisome proliferator-activated receptor (PPAR)-gamma coactivator 1alpha (PGC-1alpha), mitochondrial uncoupling protein 3 (UCP3) and hexokinase II (HKII) in primary rat skeletal muscle cells is dependent on reactive oxygen species. Biochim Biophys Acta. 2006 Sep;1763(9):969-76. doi: 10.1016/j.bbamcr.2006.06.010. Epub 2006 Jul 7. PMID 16916551
- [Background] Kang C, O'Moore KM, Dickman JR, Ji LL. Exercise activation of muscle peroxisome proliferator-activated receptor-gamma coactivator-1alpha signaling is redox sensitive. Free Radic Biol Med. 2009 Nov 15;47(10):1394-400. doi: 10.1016/j.freeradbiomed.2009.08.007. Epub 2009 Aug 14. PMID 19686839
- [Background] Irrcher I, Ljubicic V, Hood DA. Interactions between ROS and AMP kinase activity in the regulation of PGC-1alpha transcription in skeletal muscle cells. Am J Physiol Cell Physiol. 2009 Jan;296(1):C116-23. doi: 10.1152/ajpcell.00267.2007. Epub 2008 Nov 12. PMID 19005163
- [Background] Sriwijitkamol A, Coletta DK, Wajcberg E, Balbontin GB, Reyna SM, Barrientes J, Eagan PA, Jenkinson CP, Cersosimo E, DeFronzo RA, Sakamoto K, Musi N. Effect of acute exercise on AMPK signaling in skeletal muscle of subjects with type 2 diabetes: a time-course and dose-response study. Diabetes. 2007 Mar;56(3):836-48. doi: 10.2337/db06-1119. PMID 17327455
- [Background] De Filippis E, Alvarez G, Berria R, Cusi K, Everman S, Meyer C, Mandarino LJ. Insulin-resistant muscle is exercise resistant: evidence for reduced response of nuclear-encoded mitochondrial genes to exercise. Am J Physiol Endocrinol Metab. 2008 Mar;294(3):E607-14. doi: 10.1152/ajpendo.00729.2007. Epub 2008 Jan 8. PMID 18182465
- [Background] Holten MK, Zacho M, Gaster M, Juel C, Wojtaszewski JF, Dela F. Strength training increases insulin-mediated glucose uptake, GLUT4 content, and insulin signaling in skeletal muscle in patients with type 2 diabetes. Diabetes. 2004 Feb;53(2):294-305. doi: 10.2337/diabetes.53.2.294. PMID 14747278
- [Background] Phielix E, Meex R, Moonen-Kornips E, Hesselink MK, Schrauwen P. Exercise training increases mitochondrial content and ex vivo mitochondrial function similarly in patients with type 2 diabetes and in control individuals. Diabetologia. 2010 Aug;53(8):1714-21. doi: 10.1007/s00125-010-1764-2. Epub 2010 Apr 27. PMID 20422397
- [Derived] Sondergard SD, Cintin I, Kuhlman AB, Morville TH, Bergmann ML, Kjaer LK, Poulsen HE, Giustarini D, Rossi R, Dela F, Helge JW, Larsen S. The effects of 3 weeks of oral glutathione supplementation on whole body insulin sensitivity in obese males with and without type 2 diabetes: a randomized trial. Appl Physiol Nutr Metab. 2021 Sep;46(9):1133-1142. doi: 10.1139/apnm-2020-1099. Epub 2021 Mar 19. PMID 33740389